CLINICAL TRIAL: NCT02248610
Title: Follow-up in Rivaroxaban Patients in Setting of Thromboembolism
Acronym: FIRST
Status: Completed | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: FIRST registry
Record Dates: First submitted 2014-09-08; First posted 2014-09-25 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2015-08

CONDITIONS: Venous Thromboembolism
Keywords: Pulmonary embolism; PE; Deep vein thrombosis; DVT; Rivaroxaban; Venous thromboembolism; Chronic thromboembolic pulmonary hypertension; Post thrombotic limb syndrome; Root cause analysis
MeSH Terms: conditions — Venous Thromboembolism; Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Rivaroxaban: All participants will be treated with rivaroxaban.
  Interventions: Other: Non-interventional study

INTERVENTIONS:
Other: Non-interventional study

SUMMARY:
In patients with acute clots (deep vein thrombosis or pulmonary embolism) the investigators will collect real world data on their short and long term outcomes. The investigators hypothesise that in patients treated from the outset with rivaroxaban that: 1. treatment will be non-inferior to treatment with conventional anticoagulants (heparins and warfarin); 2. there will be less bleeding than when patients are on conventional anticoagulants; 3. there will be a lower long-term incidence of morbidity from chronic thromboembolic pulmonary hypertension and post-thrombotic limb syndrome.

DETAILED DESCRIPTION:
United Kingdom-only prospective, non-interventional, investigator-led, multi-centre, single cohort, registry. The observation period for each patient covers the treatment period with rivaroxaban and follow up until study end. For each patient, the treating health care professional records patient demographics, medical history, signs and symptoms, diagnosis, treatment and safety parameters at an initial visit and subsequent follow-up visit(s). Data monitoring will be undertaken by the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older with an objectively verified diagnosis of DVT and/or PE and treated according to routine clinical practice with Rivaroxaban

Exclusion Criteria:

* Patients in whom follow-up is unlikely or impossible
* Patients unable to give consent
* Patients who receive heparin therapy for more than 48 hours
* Patients who receive more than one dose of warfarin
* Patients with an indication for anticoagulation other than DVT and/or PE
* All contraindications listed in the local product information (SmPC) will form part of the exclusion criteria

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-99 years with acute DVT or PE treated with rivaroxaban, patients will have not recieved bridging anticoagulation
Sampling Method: Probability Sample
Enrollment: 1343 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of long term complications | 5 years from diagnosis of index event (DVT or PE), annual follow-up
  Incidence of long term complications as composite primary end point of VTE recurrence, PTS and CTEPH in patients treated with rivaroxaban without bridging heparin therapy

SECONDARY OUTCOMES:
Incidence of major post-thrombotic complications | 5 years from diagnosis of index event (DVT or PE), annual follow-up
  Incidence (up to 5 years) of individual major sequelae (VTE recurrence, PTS and CTEPH)
Incidence of treatment-emergent bleeding rates | 5 years from diagnosis of index event (DVT or PE), annual follow-up
  Long-term treatment-emergent bleeding rates (up to 5 years).
All-cause mortality | 5 years from diagnosis of index event (DVT or PE), annual follow-up
Treatment adherence | Full duration of anticoagulation treatment (average of 6 months)
  Adherence will be measured by patient interviews with a validated questionnaire conducted during follow-up visits.
Quality of life assessment | Full duration of anticoagulation treatment (average of 6 months)
  Regular quality of life assessment in patients diagnosed with VTE, three questionnaires to be completed at time of index event, then at second and then final clinic visits.
Healthcare resource utilisation | Full duration of anticoagulation treatment (average of 6 months)
  Healthcare resource utilisation in patients treated with long-term (>12 months) anticoagulation
Incidence of other thromboembolic events | 5 years from diagnosis of index event (DVT or PE), annual follow-up
  Long-term incidence rates of other thromboembolic events (e.g. myocardial infarction and ischaemic stroke).

OTHER OUTCOMES:
Exploratory root-cause analysis of major bleeding and recurrent VTE events | 5 years from diagnosis of index event (DVT or PE), annual follow-up
Analysis of the outpatient treatment of PE | Full duration of outpatient care (every clinic visit), until discharge (average of 6 months, 3 patient visits)
  To assess outcomes with specific reference to the patient journey (outpatient, inpatient and primary care), with particular focus on outpatient treatment of PE.
Subgroup analysis of patients with evidence of long-term VTE-related morbidity | 5 years from diagnosis of index event (DVT or PE), annual follow-up
  To identify subgroups at higher risk of adverse events (AE) and/or long-term VTE-related morbidity (PTS and CTEPH).
Evaluation of rivaroxaban in under-studied groups | 5 years from diagnosis of index event (DVT or PE), annual follow-up
  To evaluate risks of rivaroxaban in patient populations for which safety information is limited or missing (eg pregnancy, breastfeeding, patients with significant organ impairment, extremes of age).

CONTACTS AND LOCATIONS:
Overall Officials: Roopen Arya, MBChB, PhD, Principal Investigator — King's College Hospital NHS Trust
Locations (4):
- United Kingdom (4):
  - Basingstoke Hospital, Basingstoke
  - Bournemouth Hospital, Bournemouth
  - Kings College Hospital NHS Foundation Trust, London
  - Salisbury Hospital, Salisbury